CLINICAL TRIAL: NCT04834037
Title: The Effect of Provision of Information and Supportive Nursing Care on Blood Gas, Vital Signs, Anxiety, Stress and Agitation Levels in COPD Patients Treated With NIV: A Randomised Controlled Trial
Brief Title: Effect of Provision of Information and Supportive Nursing Care: A Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ilknur Aydin Avci, Head of Nursing Department, Ondokuz Mayıs University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: B.30.2.ODM.0.20.08/390
Record Dates: First submitted 2021-04-05; First posted 2021-04-06 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Anxiety, Agitation, Noninvasive Ventilation, Intensive care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Anxiety Disorders; Psychomotor Agitation

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental design
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Patients in the experimental group were provided with information in addition to routine nursing care and supportive care interventions were made. The information leaflet was explained to the patients in the experimental group face to face by the researchers and the information was repeated according to the patient's needs.
  As a pre-test measure, blood gases were taken from the patients in the experimental and control groups, their vital signs were measured, their state of consciousness was evaluated, and DASS-21 (anxiety and stress sub-dimension) and RASS (agitation dimension) were practiced by face-to-face interviews with the patients. As the last test, the same measurements were made 5 days after the first measurement and before the patients were transferred to the normal service. An information pamphlet consisting of textual material about NIV treatment was developed.
  Interventions: Behavioral: Behavioral
- No intervention (No Intervention): Routine nursing care was practiced to the control group in the intensive care clinic where the patients were located.

INTERVENTIONS:
Behavioral: Behavioral — The provision of information and supportive nursing care is recommended to alleviate anxiety, stress and agitation in COPD patients treated with NIV.
  Arms: Experimental

SUMMARY:
Background: Informative and supportive nursing care is essential to reduce complications and improve outcomes in Chronic Obstructive Pulmonary Disease (COPD) patients treated with Non-Invasive Ventilation (NIV).

Objective: Aim of the study is to determine the effect of provision of information and supportive nursing care on blood gas, vital signs, anxiety, stress and agitation levels in COPD patients treated with NIV.

Research Methodology: A randomised controlled design was used between September-December 2019. The universe of the study consisted of COPD patients treated with NIV in intensive care unit in a state hospital. A total of 60 patients, composed of 30 interventions and 30 controls, were randomly included in the sample. Provision of information and supportive nursing care was applied to the patients in the intervention group. The data were evaluated with SPSS program.

Results: Following the intervention, the findings showed that the provision of information and supportive nursing care has a positive effect on the blood gas, vital signs, anxiety, stress and agitation levels of patients.

Conclusions: The provision of information and supportive nursing care is recommended to alleviate anxiety, stress and agitation in COPD patients treated with NIV

DETAILED DESCRIPTION:
Trial design and the participants A randomised controlled design was used between September-December 2019. This study has been approved (B.30.2.ODM.0.20.08/390) by an ethics committee. In order to carry out the study, an application permit (17186359-604.02) was obtained from the Provincial Health Directorate and the relevant hospital. In addition, written consent forms were obtained from all the patients.

The sample size was determined using G * Power 3.1 software since there was no pilot data. According to the power analysis, the number of the participants was calculated as at least 54 when a type 1 error was taken as 0.05, power as 0.95, and the effect size as moderate (0.25) for two groups design with two repeated measures. In order to prevent possible data loss, the volume of the sample was increased by 10% and the total number of the participants was determined as 60. A total of 60 COPD patients treated with NIV in intensive care unit, composed of 30 interventions and 30 controls, were randomly included in the sample. Provision of information and supportive nursing care was applied to the patients in the intervention group while the control group received routine nursing care. The inclusion criteria for participants were: (a) a diagnosis of COPD (b) treated with NIV (c) be conscious of (d) agreement to participate in the study and (e) COPD patients starting NIV therapy for the first time. Patients who were intubated and therefore unable to speak, received sedation and had a Glaskow Coma Scale score below 14 were excluded. There was no drop-out during the study.

Data collection tools Personal Information Form: The form, developed by the researchers, included questions about age, gender, educational level, marital status, smoking, information on COPD, nausea and vomiting, information on NIV use.

Depression Anxiety Stress Scale (DASS-21): The scale was first developed by Lovibond and Lovibond (1995) with 42 items and three sub-dimensions. It was later revised to 21 items in 1997. The scale is 4-point Likert type, consists of 21 items and 3 sub-dimensions (depression, anxiety, stress). The adaptation of the scale to Turkish and its validity and reliability studies were conducted. Evaluation is obtained by summing the scores given to the items it contains for each sub-dimension. Minimum 0 and maximum 21 points can be obtained in all dimensions. The subscales of the scale are Cronbach's alpha values; depression 0.81, anxiety 0.80, stress 0.75.

Richmond Agitation-Sedation Scale (RASS): RASS scale was developed by a multidisciplinary team at Virginia Common Wealth University. RASS is a 10-point scale that is evaluated using verbal stimulation followed by eye contact, which is not available in other scales. It is proven that RASS has excellent validation compared to a wide range of visual analog scales and selected sedation measurements for adult medical and surgical intensive care patients. While zero (0) points on the scale indicate the ideal level, it reflects the increasing agitation towards the (+4) level and the decreasing sedation level to the (-5) level. Since patients receiving sedation were not included in this study, only the agitation dimension of the RASS scale was used.

Glaskow Coma Scale (GCS): It was developed in Scotland / Glasgow in 1974 to describe the consciousness level of patients. The scale is widely used to assess patients' level of consciousness. There are 3 separate sections in the scale: eye opening, verbal and motor response. GCS is obtained by summing the points the patient gets from each section. This score ranges from three (3) to fifteen (15). If the GCS total score is 13-15, the patient is considered awake, between 8-12 as precoma, and below 8 as coma.

Intervention Patients in the experimental group were provided with information in addition to routine nursing care and supportive care interventions were made. The information leaflet was explained to the patients in the experimental group face to face by the researchers and the information was repeated according to the patient's needs. Supportive nursing care was also practiced to the patients in the experimental group by the researchers. Routine nursing care was practiced to the control group in the intensive care clinic where the patients were located.

As a pre-test measure, blood gases were taken from the patients in the experimental and control groups, their vital signs were measured, their state of consciousness was evaluated, and DASS-21 (anxiety and stress sub-dimension) and RASS (agitation dimension) were practiced by face-to-face interviews with the patients. As the last test, the same measurements were made 5 days after the first measurement and before the patients were transferred to the normal service.

An information pamphlet consisting of textual material about NIV treatment was developed. The content of the information leaflet consisted of topics that will facilitate patient compliance to treatment, such as the introduction of equipment used in NIV treatment, the intended use of NIV and its effects on the patient, what patients generally experience during treatment, compliance problems in NIV, how the procedure will be performed, each procedure the nurse will do and for what purpose, the duration of the treatment, what the patient can and cannot do during the treatment, what kind of process will proceed if everything goes well. As supportive care, patients were allowed to express their feelings and thoughts about NIV treatment, an accepting and empathetic approach was shown to the patients, care was taken to make eye contact while communicating, therapeutic touch technique was used, it was explained how the patients could reach the nurse when needed, the environment was arranged, each procedure performed was explained with its objectives, they were placed in a position where they could see the clock, strategies that will make it easier for the patients to cope during the treatment were determined and they were encouraged to do so (for example, some patients wanted to read a book and some patients wanted to sleep), the patients were encouraged to ask questions comfortably, it was stated that the treatment could be interrupted for a while when they felt bad due to the mask, and it was ensured that the patients met with their relatives during the visiting hours.

Data analysis The Statistical Package for Social Sciences (SPSS) 20.0 package program was used in the analysis of the data. Descriptive statistics were used as mean ± standard deviation for variables with normal distribution, and median (min - max) for variables with non-normal distribution. Nominal variables were shown as the number of patients (n) and (%). The compliance of the data to normal distribution was examined with the Shapiro-Wilk test and the homogeneity of the variances with the Levene test. For the comparison of the experimental and control groups, Student's T test was used for data with normal distribution, Mann Whitney U test was used for data with non-normal distribution. Chi-Square and Fisher's Exact tests were used for group comparisons of nominal variables. "Analysis of Variance in Repeated Measures" was used to analyze the values of the experimental and control groups before and after the training in order to evaluate the effectiveness of the provision of information and supportive nursing care intervention practised to the experimental group. In the analysis of all tests, p value <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of COPD treated with NIV be conscious of agreement to participate in the study COPD patients starting NIV therapy for the first time

Exclusion Criteria:

* intubated therefore unable to speak received sedation had a Glaskow Coma Scale score below 14 were excluded

Ages: 48 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Depression Anxiety Stress Scale (DASS-21) | 3 months
  The scale was first developed by Lovibond and Lovibond (1995) with 42 items and three sub-dimensions. It was later revised to 21 items by Brown et al. (1997) in 1997. The scale is 4-point Likert type, consists of 21 items and 3 sub-dimensions (depression, anxiety, stress). The adaptation of the scale to Turkish and its validity and reliability studies were conducted by Yılmaz et al. (2017). Evaluation is obtained by summing the scores given to the items it contains for each sub-dimension. Minimum 0 and maximum 21 points can be obtained in all dimensions. The subscales of the scale are Cronbach's alpha values; depression 0.81, anxiety 0.80, stress 0.75 (Yılmaz et al., 2017).
Richmond Agitation-Sedation Scale (RASS) | 3 months
  RASS scale was developed by a multidisciplinary team at Virginia Common Wealth University (Sessler et al. , 2002). RASS is a 10-point scale that is evaluated using verbal stimulation followed by eye contact, which is not available in other scales. It is proven that RASS has excellent validation compared to a wide range of visual analog scales and selected sedation measurements for adult medical and surgical intensive care patients. While zero (0) points on the scale indicate the ideal level, it reflects the increasing agitation towards the (+4) level and the decreasing sedation level to the (-5) level. Since patients receiving sedation were not included in this study, only the agitation dimension of the RASS scale was used.
Glaskow Coma Scale (GCS) | 3 months
  It was developed in Scotland / Glasgow in 1974 to describe the consciousness level of patients. The scale is widely used to assess patients' level of consciousness. There are 3 separate sections in the scale: eye opening, verbal and motor response. GCS is obtained by summing the points the patient gets from each section. This score ranges from three (3) to fifteen (15). If the GCS total score is 13-15, the patient is considered awake, between 8-12 as precoma, and below 8 as coma (Sepit, 2005).

CONTACTS AND LOCATIONS:
Overall Officials: İlknur AYDIN AVCİ, Prof., Study Director — Ondokuz Mayıs University; Yasemin ÇEKİÇ, Dr., Principal Investigator — Ankara University; Tuba YILMAZ BULUT, Msc, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Bafra State Hospital, Samsun, Turkey (Türkiye)